CLINICAL TRIAL: NCT02773550
Title: Clinical, Multicenter, Single-arm, Treatment With a Scheme With Low Doses of Bortezomib / Melphalan / Prednisone (MPV) in Patients With Multiple Myeloma (MM) Newly Diagnosed Symptomatic ≥75 Years
Brief Title: Treatment With a Scheme With Low Doses of Bortezomib / Melphalan / Prednisone (MPV) in Patients With Multiple Myeloma
Acronym: Velcadito
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruiment.
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Ernesto Perez Persona, Doctor, Basque Health Service
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Velcadito
Record Dates: First submitted 2015-03-25; First posted 2016-05-16 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2016-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Velcadito (Experimental): Bortezomib 1.3 mg/m2 days 1,4,8 and 11 first cycle, the 1.0 mg/m2 days 1 and 4. Melphalan 9 mg/m2 days 1 to 4 Prednisone 60 mg/m2 days 1 to 4 Cycles of 28 days
  Interventions: Drug: Bortezomib; Drug: Melphalan; Drug: Prednisone

INTERVENTIONS:
Drug: Bortezomib — Low dose of bortezomib
  Other Names: Velcade
Drug: Melphalan
Drug: Prednisone

SUMMARY:
This clinical trial is a multicenter, cohort, with one arm to study the SLP to 18 months of Velcadito scheme (velcade 1.0 mg / m2 administered over two days with melphalan and prednisone) in patients with MM diagnosis again higher 75. After completion of the protocol patients were still approximately every two months, in clinical practice, to observe the survival and answers to other treatments. All the scans are part of the normal routine. The realization of diagnostic tests and drug treatment will be performed regardless of the patient's participation in the study as part of routine clinical practice All patients who meet criteria. The incidence of MM age-adjusted to cover the participating hospitals is estimated in 44 patients.

Patients will receive a course of 4 weeks duration of Melphalan / Prednisone / Velcade consist in Melphalan, 9 mg / m2 orally daily 1-4 and Prednisone 60 mg / m2 orally on days 1 to 4, in combination Velcade with a dose of 1.3 mg / m2 sc twice weekly (days 1, 4, 8, 11), followed by 2 weeks of rest (cycle duration of 4 weeks) and seven four-week cycles duration of melphalan / prednisone / Velcade consist in Melphalan, 9 mg / m2 orally on days 1 to 4 and prednisone, 60 mg / m2 orally on days 1 to 4, in combination with Velcade, at doses of 1, 0 mg / m2 sc (days 1, 4).

Melphalan and Prednisone will be dispensed for oral administration. The Melphalan should be administered in a single two hours separately taking any food and prednisone be taken in the morning with or immediately after a meal. The amount in mg will be calculated based on the body surface, to be calculated on day 1 of each cycle. Velcade for administration, calculated on day 1 of the cycle will be the same dose throughout the entire cycle. If a patient experiences a gain or loss of remarkable weight within the cycle, the dose to be administered will be recalculated based on the new body surface. The appropriate amount of Velcadeserá dispensed in a sc injection. Velcade dose between two leave at least 72 hours

DETAILED DESCRIPTION:
This clinical trial is a multicenter, cohort, with one arm to study the SLP to 18 months of Velcadito scheme (velcade 1.0 mg / m2 administered over two days with melphalan and prednisone) in patients with MM diagnosis again higher 75. After completion of the protocol patients were still approximately every two months, in clinical practice, to observe the survival and answers to other treatments. All the scans are part of the normal routine. The realization of diagnostic tests and drug treatment will be performed regardless of the patient's participation in the study as part of routine clinical practice All patients who meet criteria. The incidence of MM age-adjusted to cover the participating hospitals is estimated in 44 patients.

Clinical Study Materials:

* Melphalan is presented for oral administration of 2 mg tablets.
* Prednisone is presented for oral administration in tablets 50, 30, 10, 5 and 2.5 mg to set the correct dose to be administered.
* Velcade.- (Bortezomib) for subcutaneous administration. All study drugs will be administered to patients under the prescription of the investigator or sub-investigators identified and in the case of Velcade dispensed in hospital Pharmacy Service Patients will receive a course of 4 weeks duration of Melphalan / Prednisone / Velcade consist in Melphalan, 9 mg / m2 orally daily 1-4 and Prednisone 60 mg / m2 orally on days 1 to 4, in combination Velcade with a dose of 1.3 mg / m2 sc twice weekly (days 1, 4, 8, 11), followed by 2 weeks of rest (cycle duration of 4 weeks) and seven four-week cycles duration of melphalan / prednisone / Velcade consist in Melphalan, 9 mg / m2 orally on days 1 to 4 and prednisone, 60 mg / m2 orally on days 1 to 4, in combination with Velcade, at doses of 1, 0 mg / m2 sc (days 1, 4).

Melphalan and Prednisone will be dispensed for oral administration. The Melphalan should be administered in a single two hours separately taking any food and prednisone be taken in the morning with or immediately after a meal. The amount in mg will be calculated based on the body surface, to be calculated on day 1 of each cycle. Velcade for administration, calculated on day 1 of the cycle will be the same dose throughout the entire cycle. If a patient experiences a gain or loss of remarkable weight within the cycle, the dose to be administered will be recalculated based on the new body surface. The appropriate amount of Velcadeserá dispensed in a sc injection. Velcade dose between two leave at least 72 hours

ELIGIBILITY:
Inclusion Criteria:

* The patient should, in the investigator's opinion, be able to meet all requirements of the trial.
* The patient must voluntarily sign informed consent before performing any test study that is not part of routine care of patients, with the knowledge that the patient can leave the study at the time you want, without being harmed at any time their aftercare.
* Age > 75 years.
* The patient should be diagnosed symptomatic multiple myeloma according to established criteria and may not have received any treatment for disease (see Appendix 6). Administration is permitted steroid pulses some urgency required prior to starting treatment or induction administration of bisphosphonates.

The patient must have measurable disease, defined as follows:

* For Multiple Myeloma secretory measurable disease is defined by the presence of measurable serum monoclonal component, 1g/dL or if urinary excretion of light chains is greater than or equal to 200 mg/24 hours.
* For Multiple Myeloma oligosecretory or secretory, serous level chain.
* Free light affected 10 mg/dL (100 mg/L, with a ratio of abnormal free light chain serum).
* The patient must have a life expectancy greater than 3 months life.
* The patient must have the following laboratory values prior to initiation of treatment corresponding induction:

  * Platelet count 50000/mm3,
  * hemoglobin 8 g/dl,
  * absolute neutrophil count 1000/mm3,
  * Lower values are permitted if they are due to infiltration of the MO.

Exclusion Criteria:

* Patients who have previously received treatment for multiple myeloma, with the exception of steroid pulses for some urgency required prior to initiating induction therapy, administration of bisphosphonates or radiotherapy either analgesic or due to the presence of plasmacytomas require it for some urgency.
* Patients with non-measurable disease or by SFLC.
* Patients with known hypersensitivity to bortezomib, boron or mannitol acid.
* Patients who have received any investigational agent within 30 days prior to enrollment.
* Patients who are currently in another clinical trial or receiving any investigational agent.
* Hypertension or poorly controlled diabetes mellitus or other serious organic disease involving excessive risk to the patient or any psychiatric disorder that interfere with the understanding of informed consent.
* Acute diffuse infiltrative pulmonary disease and pericardial disease.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Pérez Persona, Study Director — Hospital Universitario Araba (Sede Txogoriritxu)
Locations (1):
- Araba of University Hospital, Vitoria-Gasteiz, Araba, Spain

IPD SHARING:
Plan to Share IPD: No